CLINICAL TRIAL: NCT05551221
Title: The Efficacy and Safety of Silodosin Singly or Combined With Ningmitai Capsules in the Treatment of Benign Prostatic Hyperplasia (BPH) Complicated With Lower Urinary Tract Symptoms (LUTS) -A Multicenter, Prospective, Randomized, Double-blind, Positive Controlled Study
Brief Title: The Efficacy and Safety of Silodosin Singly or Combined With Ningmitai Capsules in the Treatment of Benign Prostatic Hyperplasia
Acronym: NQTIPS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREC2022-17
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Benign Prostatic Hyperplasia With Lower Urinary Tract Symptoms
Keywords: Benign Prostatic Hyperplasia Silodosin Capsules; Ningmitai Capsule; Silodosin
MeSH Terms: interventions — silodosin; Tamsulosin

STUDY DESIGN:
Intervention Model Description: Group A: Oral Tamsulosin Hydrochloride Capsules and Ningmitai Capsules placebo for 12 weeks.
  Group B: Oral l Silodosin Capsules and Ningmitai Capsules placebo for 12 weeks. Group C: Oral l Silodosin Capsules and Ningmitai Capsules for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tamsulosin Hydrochloride Capsules combine with Ningmitai Capsules placebo (Active Comparator): Patients take tamsulosin hydrochloride capsules (1 tablet each time, once daily) and Ningmitai capsules placebo (0.38 g/capsule, 4 capsules/time, tid.)
  Interventions: Drug: Tamsulosin
- Silodosin Capsules combine with Ningmitai Capsules placebo (Experimental): Patients take Silodosin Capsules ( Qianweitai®, 4mg/capsule, 1 capsule/time, bid, after breakfast and dinner) and Ningmitai capsules placebo (0.38 g/capsule, 4 capsules/time, tid).
  Interventions: Drug: Silodosin Capsules
- Silodosin Capsules combine with Ningmitai Capsules (Experimental): Patients take Silodosin Capsules ( Qianweitai®, 4mg/capsule, 1 capsule/time, bid, after breakfast and dinner) and Ningmitai capsules (Ningmitai®, 0.38 g/capsule, 4 capsules/time, tid).
  Interventions: Drug: Silodosin Capsules; Drug: Ningmitai capsule

INTERVENTIONS:
Drug: Silodosin Capsules — Silodosin is a α1A-adrenergic receptor antagonist which can relax the smooth muscle of bladder and prostate, relieves the dynamic obstruction of bladder outlet, and improves the lower urinary tract symptoms caused by BPH. The instruction of Silodosin Capsule (Qianweitai®) is 4mg/capsule，1 capsule/time, bid, after breakfast and dinner.
  Other Names: Qianweitai
  Arms: Silodosin Capsules combine with Ningmitai Capsules; Silodosin Capsules combine with Ningmitai Capsules placebo
Drug: Ningmitai capsule — Ningmitai Capsule (Ningmitai®) is Traditional Chinese Medicine which has already used in treatment of urinary system disease (eg. CPPS, BPH) in China for more than twenty years. The instruction of Ningmitai Capsule is 0.38g/capsule, 4 capsule/time, tid.
  Other Names: Ningmitai
  Arms: Silodosin Capsules combine with Ningmitai Capsules
Drug: Tamsulosin — Tamsulosin is α1A-adrenergic receptor which has used in treatment of BPH for few years. The instruction of Tamsulosin Capsule is 1 tablet at a time, 1 time a day.
  Arms: Tamsulosin Hydrochloride Capsules combine with Ningmitai Capsules placebo

SUMMARY:
Objective: To evaluate the efficacy and safety of Ningmitai Capsules and Silodosin Capsules in the treatment of Benign Prostatic Hyperplasia (BPH) with Lower Urinary Tract Symptoms (LUTS) compared with Tamsulosin Hydrochloride Sustained Release Capsules.

Study design: A multicenter, prospective, randomized, double-blind, positive controlled clinical study.

Interventions:

Group A: Oral Tamsulosin Hydrochloride Capsules and Ningmitai Capsules placebo for 12 weeks.

Group B: Oral l Silodosin Capsules and Ningmitai Capsules placebo for 12 weeks. Group C: Oral l Silodosin Capsules and Ningmitai Capsules for 12 weeks.

DETAILED DESCRIPTION:
Sample size: 312

ELIGIBILITY:
Inclusion Criteria:

1. Male Subjects aged 60 ～ 80 years, clinically diagnosed as benign prostatic hyperplasia.
2. Has an IPSS score ≥ 8 points at Screening and Baseline.
3. Has a 4 ≤ Qmax ≤ 15 ml/s when urination volume > 150 ml.
4. Has a prostate volume (PV) ≥ 30 ml by ultrasound examination.
5. Subjects who can read, understand, and complete the research questionnaire.
6. Subjects willing to participate voluntarily in this clinical trial, give informed consent and sign informed consent.

Exclusion Criteria:

1. Subjects with prostate cancer or other malignant tumors.
2. Subjects have serum tPSA > 10ng/ml, or 4 ≤ tPSA ≤ 10ng/ml while fPSA/tPSA < 0.16 times.
3. Subjects suffered from other diseases causing dysuria, such as bladder neck spasm, urethral stricture, neurogenic bladder dysfunction, etc.
4. Subjects have suffered from acute urinary retention, or complicated with gross hematuria, urinary tract infection, bladder stones, secondary upper urinary tract hydronephrosis, urinary incontinence, renal insufficiency and other Subjects that researchers believe meet the surgical indications.
5. Subjects have undergone prostate surgery, microwave therapy, urethral dilatation or acute urinary retention catheterization or other invasive procedures.
6. Subjects have residual urine volume (PVR) > 100ml, or those who may have urinary retention and need catheterization.
7. Subjects who took α receptor blockers, traditional Chinese medicine or botanical drugs for treating BPH within two weeks before participating this clinical trial.
8. Subjects who take 5α reductase inhibitor or other antiandrogen therapy drugs within half a year before participating this clinical trial.
9. Subjects who need to take drugs prohibited in this study or adopt prohibited treatment methods during treatment.
10. Subjects who Complicated with severe cardiovascular and cerebrovascular diseases, respiratory diseases, blood diseases, liver and kidney diseases.
11. There are significant abnormalities in clinical or laboratory examination indexes of patients, such as ALT and AST ≥ 2.5 times of the upper limit of reference value, creatinine (Scr) > 1.5 times of the upper limit of reference value, or poor blood glucose control (fasting blood glucose FPG ≥ 10 mmol/L).
12. Subjects who are allergic to the drugs or ingredients used in the test definitely.
13. Any otherSubjects in the opinion of researchers is not suitable for inclusion.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score（IPSS） | 12 week
  Changes of IPSS scores at the 12th week of treatment compared with baseline scores. The scores of the scale ranged from 0 to 35. The higher the score, the more severe the symptoms are.

SECONDARY OUTCOMES:
International Prostate Symptom Score（IPSS） total score | 1, 2, 4 and 8 weeks
  Changes of IPSS scores at 1, 2, 4 and 8 weeks after treatment compared with baseline scores. The scores of the scale ranged from 0 to 35. The higher the score, the more severe the symptoms are.
IPSS Stimulus score | 1, 2, 4 ,8 and 12 weeks
  IPSS Stimulation Score at 1, 2, 4, 8, 12 weeks (Sum of Question 2, 4, 7) compared with baseline. The scores of the scale ranged from 0 to 15. The higher the score, the more severe the symptoms are.
IPSS obstruction score | 1, 2, 4 ,8 and 12 weeks
  Changes of IPSS obstruction score (sum of question 1, 3, 5, 6) at 1, 2, 4, 8, 12 weeks after treatment compared with baseline. The scores of the scale ranged from 0 to 20. The higher the score, the more severe the symptoms are.
IPSS total score severity | 12 week
  Proportion of patients with IPSS total score severity decreased by at least one grade at 12 weeks. The scores of the scale were divided into three grades: mild (0-7), moderate (8-19) and severe (20-35).
Quality of life (QoL) score | 4, 8 and 12 weeks
  Changes in scores at 4, 8 and 12 weeks of treatment compared with baseline.The scores of the scale ranged from 0 to 6. The higher the score, the more severe the symptoms are.
Maximum urinary flow rate (Qmax) | 12 weeks
  The change of Qmax at 12 weeks of treatment compared with baseline.
Residual urine volume (PVR) | 12 weeks
  Changes of PVR at 12 weeks of treatment compared with baseline.
Prostate specific antigen (PSA) | 12 weeks
  Changes of PSA at 12 weeks of treatment compared with baseline.
Prostate volume (PV) | 12 weeks
  Changes of PV at 12 weeks of treatment compared with baseline.
Patient response rate | 12 weeks
  Patient response rate is defined as the proportion of patients whose IPSS total score decreased by ≥ 25% and Qmax increased by ≥ 30% compared with baseline value after treatment.
Proportion of patients with BPH clinical progression | 12 weeks
  Clinical progress is defined as the first occurrence of one of the following two conditions during the trial:
  1. Acute urinary retention (AUR);
  2. Clinical diagnosis requires surgical treatment of BPH.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongguo Chen, MD, Study Chair — employee
Locations (8):
- China (8):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Central Hospital Of WUHAN, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05551221/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05551221/SAP_001.pdf